CLINICAL TRIAL: NCT02606448
Title: Liposomal Bupivacaine Versus Femoral Nerve Block for Pain Control After Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Trial
Brief Title: Exparel Infiltration in Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Sub Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXP-ACL
Record Dates: First submitted 2015-10-05; First posted 2015-11-17 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Pain
Keywords: pain control; patient satisfaction; liposomal bupivacaine; Anterior cruciate ligament reconstruction
MeSH Terms: conditions — Pain; Agnosia; Patient Satisfaction | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femoral Nerve Block (Active Comparator): Patients in this group received preoperative ultrasound guided femoral nerve blocks by senior anesthesiologist using ropivicaine.
  Interventions: Procedure: Femoral nerve block; Drug: Ropivacaine
- Liposomal Bupivacaine (Experimental): Patients in this group received local infiltration of Liposomal bupivacaine before the end of surgery.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Local infiltration of liposomal bupivacaine
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Procedure: Femoral nerve block — Pre-operative femoral nerve block
  Arms: Femoral Nerve Block
Drug: Ropivacaine — Ropivicaine was used in all femoral nerve blocks
  Arms: Femoral Nerve Block

SUMMARY:
This is a randomized, single blinded, standard of care controlled clinical trial. All adult patients over sixteen desiring anterior cruciate ligament reconstruction will be eligible. The study compares pain control and opioid consumption in patients undergoing ACL reconstruction between patients receiving liposomal bupivacaine and those who underwent a preoperative femoral nerve block.

DETAILED DESCRIPTION:
Study Design: A randomized single blinded standard of care controlled clinical trial comparing pain management interventions. All patients over age sixteen and scheduled for primary or revision anterior cruciate ligament reconstruction (ACL) a single fellowship trained sports surgeons will be eligible for inclusion. Patients will be excluded if their medical history presents known allergies or intolerance to dexamethasone, opioid or bupivacaine, substantial alcohol or drug abuse, and pregnancy. Secondary exclusion criterion is an intact ACL.

Liposomal Bupivacaine has a refrigerated shelf life of one month in our facility. Patients will be sequentially recruited into the randomization process. Liposomal Bupivacaine will be held by the Henry Ford hospital pharmacy up to one month prior to planned anterior cruciate ligament reconstruction in anticipation of surgery on eligible patients. The sterile solutions will be delivered to and kept by the inpatient clinical pharmacy until the date of surgery and delivered to the operating room at the beginning of a surgical case. The current dose of Liposomal Bupivacaine has been chosen based on previously published data of local infiltrative analgesia with Liposomal Bupivacaine and one published study on Liposomal Bupivacaine efficacy.

The week prior to surgery, patients will be randomized to receive Local infiltration anesthesia (LIA) with Liposomal Bupivacaine, or Femoral nerve block (FNB) using a computer generated sequence. The results of randomization will be securely delivered to the anesthesiologist and the surgeon the week prior. The anesthesiologist will view the assigned group to determine if a preoperative FNB will be given. Depending on the randomization group either an Liposomal Bupivacaine solution will be delivered to the operating room for local infiltration or the anesthesiologist will perform a preoperative FNB.

Patients in the Liposomal Bupivacaine group will receive LIA with 10cc(133mg) of Liposomal Bupivacaine solution dissolved in 20cc of sterile saline after harvest of the hamstring graft or patella tendon graft. The solution will be applied to the wound bed, graft site, and periosteum. The solution will be left unperturbed for five minutes. Thereafter the solution will be suctioned from the wound and the knee joint. Incisions will be closed in typical fashion and the wound dressed.The tourniquet will be deflated.

Patient in the FNB will receive postoperative ultrasound guided FNB. Experienced anesthesiologists will apply all FNBs in this study.

Following the procedure pain will be accessed subjectively through visual analog scale and numeric rating scale pain scores, pain diaries given to the patient to record at home, pain summary scores at follow up visits and objectively through narcotic pain requirement. A blind observer will also access outcomes.

Planned Data Analysis:

Means and standard deviations, as well as medians and interquartile ranges will be computed for pain scores.These outcomes will be compared by Wilcoxon rank sum tests. The amount of pain medication and pain scores will be compared by Wilcoxon rank sum tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 16 scheduled for primary or revision anterior cruciate ligament reconstruction by one fellowship trained sports surgeon will be eligible for inclusion

Exclusion Criteria:

* Patients will be excluded if their medical history presents known allergies or intolerance to dexamethasone, opioid or bupivacaine, substantial alcohol or drug abuse, and pregnancy. Secondary exclusion criterion is an intact ACL

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pain levels | 4 days postoperatively
  Patients recorded pain lvls every four hours using VAS scales for four days post operatively

SECONDARY OUTCOMES:
Morphine equivalents | 4 days postoperatively
  Patients recorded opioid intake for four days postoperatively